CLINICAL TRIAL: NCT06066476
Title: A Prospective, Multicenter, Observational Study to Evaluate the Efficacy and Safety of GENOSS DES in Patients with Coronary Artery Disease
Brief Title: Efficacy and Safety of GENOSS® DES in Patients with Coronary Artery Disease
Acronym: GENOSSRegistry
Status: Completed | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-DS0501-08
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GENOSS Sirolimus Eluting Coronary Stent System: Patients with coronary artery disease treated with the GENOSS DES

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of the GENOSS DES in patients with coronary artery disease in real-world pratice.

DETAILED DESCRIPTION:
The Genoss DES is a novel, biodegradable, polymer-coated, sirolimus-eluting stent with a cobalt-chromium stent platform and thin strut. Although the efficacy and safety of this stent have been previously investigated, real-world clinical outcomes data are lacking. Therefore, the objective of this prospective, multicenter study was to evaluate the clinical efficacy and safety of the Genoss DES in all-comer patients undergoing percutaneous coronary intervention.

The Genoss DES registry is a prospective, single-arm, observational study for evaluation of clinical outcomes after Genoss DES implantation in all-comer patients undergoing percutaneous coronary intervention from 12 sites in South Korea. The primary endpoint was a device-oriented composite endpoint (DOCE), defined as a composite of cardiac death, target vessel-related myocardial infarction (MI), and clinically indicated target lesion revascularization (TLR) at 12 months.

ELIGIBILITY:
<Inclusion Criteria>

1. Patients of 19 and over
2. Patients eligible for treatment of coronary artery disease using GENOSSTM DES
3. Participants who voluntarily decide to participate in this clinical trial, agree to the study protocol and clinical follow-up plan, and provide written informed consent as research participants.

<Exclusion Criteria>

1. Patients who are contraindicated in the use of heparin, aspirin, clopidogrel, sirolimus, cobalt chromium and contrast agents (However, patients with hypersensitivity to contrast agents may be eligible if it can be controlled by steroids and pheniramine. Patients with known anaphylaxis are excluded)
2. Patients who are pregnant or planning to become pregnant
3. Patients scheduled to undergo surgery requiring the discontinuation of antiplatelet agents within 12 months from registration
4. Patients with a life expectancy of less than 1 year
5. Patients who presented with cardiogenic shock at admission and are predicted to have a low chance of survival based on medical judgment
6. Patients who have already received treatment with another DES (Drug Eluting Stent), BVS (Bioresorbable Vascular Scaffolds), or BMS (Bare Metal Stent) at the time of registration
7. Patients currently participating in a randomized controlled trial involving medical devices

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease treated with GENOSS DES
Sampling Method: Non-Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2017-06-24 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Device-oriented composite endpoint | at 12 months after the procedure
  DOCE is defined as a composite of cardiac death, target vessel-related myocardial infarction (TV-MI) and clinically indicated target-lesion revascularization (TLR).

SECONDARY OUTCOMES:
Patient-oriented composite endpoint | at 12 months after the procedure
  POCE is defined as a composite of all-cause death, any myocardial infarction, and any revascularization.
All-cause deaths | at 12 months after the procedure
Cardiac death | at 12 months after the procedure
Non-cardiac death | at 12 months after the procedure
Any myocardial infarction | at 12 months after the procedure
target vessel-related myocardial infarction (TV-MI) | at 12 months after the procedure
Any revascularization | at 12 months after the procedure
Clinically indicated target lesion revascularization (TLR) | at 12 months after the procedure
Stent thrombosis | at 12 months after the procedure
Lesion success | during the procedure
  When the final residual lesion stenosis is less than 50% using any surgical method.
Procedure success | immediately after the procedure
  When the final residual lesion stenosis is less than 50% using any surgical method, and there is no post-procedure death, myocardial infarction, or revascularization during the hospitalization period.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The data set is available from the the corresponding author upon reasonable request.